CLINICAL TRIAL: NCT07143331
Title: A Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetic Profile of Single and Multiple Ascending Doses of KS101 in Healthy Volunteers, Including a Pilot Food Effect Evaluation
Brief Title: A Phase 1 Study to Assess the Safety and Effects of Single and Multiple Doses of KS101 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Klotho Sciences Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Organization: Klotho Sciences (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: KS101-CLIN-001
Record Dates: First submitted 2025-08-03; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants; Alzheimer Disease; Chronic Kidney Disease
Keywords: alzheimer disease; chronic kidney disease
MeSH Terms: conditions — Alzheimer Disease; Renal Insufficiency, Chronic | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1 KS101 (Experimental): Participants will be enrolled in 1 of 6 single ascending dose cohorts. Six participants in each cohort will receive KS101.
  Interventions: Drug: Part 1 KS101
- Part 1 Placebo (Placebo Comparator): 6 doses of placebo will be administered to participants
  Interventions: Drug: Part 1 Placebo
- Part 2 KS101 with Food (Experimental): KS101 with food
  Interventions: Drug: Part 2 with Food
- Part 2 KS101 without Food (Experimental): KS101 without food
  Interventions: Drug: Part 2 without food
- Part 3 KS101 (Experimental): Multiple ascending doses of KS101
  Interventions: Drug: Part 3 KS101

INTERVENTIONS:
Drug: Part 1 KS101 — Six doses of oral KS101 will be administered to participants.
  Arms: Part 1 KS101
Drug: Part 1 Placebo — Six doses of oral matching placebo will be administered to participants.
  Arms: Part 1 Placebo
Drug: Part 2 with Food — KS101 administered with food
  Arms: Part 2 KS101 with Food
Drug: Part 2 without food — KS101 administered without food
  Arms: Part 2 KS101 without Food
Drug: Part 3 KS101 — 3 multiple doses of KS101
  Arms: Part 3 KS101

SUMMARY:
This study is the first clinical trial involving study drug KS101. The goal of this clinical trial is to investigate whether KS101 is safe, whether it causes side effects, and how KS101 is broken down in the body, in healthy participants.

This information will be used to learn more about KS101 and to determine the most effective dose for age related diseases such as chronic kidney disease and Alzheimer's Disease, with the fewest unwanted side effects.

There are 3 parts to this study. In Part 1, participants will take KS101 or a placebo once and will stay in the study centre for a 4-night inpatient stay. Participants will return for outpatient visits on Days 8 and 29.

In Part 2, participants will take KS101 twice, once after a meal and once without a meal and will stay in the study centre for a 7-night inpatient stay. Participants will return for outpatient visits on Days 11 and 32.

In Part 3, participants will take KS101 or a placebo once daily for 5 days and will stay in the study centre for an 8-night inpatient stay. Participants will return for outpatient visits on Days 12 and 33.

DETAILED DESCRIPTION:
This is a Phase 1, 3-part study to evaluate the safety, tolerability, and pharmacokinetic (PK) profile following the oral administration of single and multiple ascending doses of KS101 in healthy participants, including a food effect evaluation.

Part 1 will include six single ascending dose cohorts of 8 participants per cohort (randomised 6 active, 2 placebo). For each cohort, a sentinel group of 2 participants (1 active, 1 placebo) will be dosed first. These participants will be on study for up to 59 days in total.

Part 2 will be a crossover evaluation, with and without food (randomised sequence). 12 participants will receive 2 doses of KS101 72 hours apart, one dose under fasting conditions and one dose under fed conditions. These participants will be on study for up to 61days in total.

Part 3 will include three multiple ascending dose cohorts of 8 participants per cohort (randomised 6 active, 2 placebo). These participants will receive one dose for 5 consecutive days and will be on study for up to 63 days in total.

ELIGIBILITY:
Inclusion Criteria:

1. Provided voluntary, written informed consent before any study-specific activities are performed.
2. Male or female, aged 18 to 55 years inclusive at time of informed consent.
3. Participants of childbearing potential must agree to the use of a double method of contraception of a highly effective method of birth control (refer to Appendix 11.1) combined with a barrier contraceptive (condom) when appropriate from screening visit to until 60 days after the last dose of IMP (covering a full menstrual cycle of 30 days starting after 5 half-lives of last dose of IMP). Childbearing potential is defined as fertile and following menarche until becoming post-menopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Post-menopausal is defined as no menses for 12 months without an alternative medical cause and a Screening follicle stimulating hormone (FSH) level >30 U/L (or at the local laboratory levels for post-menopause).
4. Male participants with sexual partners of childbearing potential must agree to use a double method of contraception including condom with a highly effective method of birth control by the partner of childbearing potential (refer to Appendix 11.1), from the time of informed consent through to 90 days after the last dose of the IMP. Male participants who have undergone sterilisation (i.e., vasectomy ≥6 months before Screening) and have had testing to confirm the success of the sterilisation, may also be included and will not be required to use above described methods of contraception. Male participants must also agree not to donate sperm or plan to father children for up to 90 days after last dose of IMP.
5. Non-smoker (or other nicotine use) (defined as ≤5 cigarettes or nicotine equivalent per month) for at least 32 months before Screening according to history, and urine cotinine <500 ng/mL or carbon monoxide (CO) breath test <10 ppm at Screening and Day -1.
6. Total body weight ≥50 kg (male) or ≥45 kg (female) and body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive.
7. Certified as healthy by comprehensive clinical assessment by the Investigator (detailed medical history, complete physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory evaluation) and with suitable veins for cannulation.
8. Vital signs after 5 minutes resting in supine position (one repeat per timepoint permitted):

   * Systolic blood pressure (SBP): 90 - 140 mmHg inclusive
   * Diastolic blood pressure (DBP): 50 - 90 mmHg inclusive. DBP 40 - 49 mmHg inclusive is acceptable for eligibility if considered not clinically significant by the Investigator.
   * Heart rate (HR): 50 - 90 bpm inclusive. HR 40 - 49 bpm inclusive are acceptable for eligibility if considered not clinically significant by the Investigator.
9. Standard 12-lead electrocardiogram (ECG) parameters, after 10 minutes in supine position within the following ranges:

   * QRS 50 - 120 msec
   * QT ≤500 msec
   * QTcF and QTcB ≤450 msec (male) ≤470 msec (female) Also: normal ECG tracing, or ECG tracing abnormality considered by the Investigator to be not clinically significant (not including parameters above).
10. In the opinion of the Investigator, is willing and able to comply with and understand study requirements provided in English and be available for the required study visits. For Part 2 FE, this includes being willing and able to consume a high-fat meal (≥50% fat) within 30 minutes.
11. Is willing to defer blood donations to a blood service for minimum 6 months after the End of study visit.

Exclusion Criteria:

1. Liver function tests at Screening and Day -1: aspartate aminotransferase [AST], alanine aminotransferase [ALT],) >2 times upper limit of normal (ULN), serum alkaline phosphatase (ALP) or total bilirubin ≥2 times ULN. One re-test per parameter per timepoint is permitted, results must be available before randomization.
2. Clinically significant abnormalities in laboratory tests (biochemistry, haematology, coagulation, urinalysis), physical examination, or 12-lead ECG during the Screening period or pre-first dose, that in the opinion of the Investigator, would affect the individual's ability to fully participate in the study and/or not be in the individual's best interest to participate in the study. One re-test per abnormality per scheduled timepoint is permitted
3. Pregnant or breastfeeding, or planning to become pregnant or breastfeed, or planning to donate ova during study participation; or positive pregnancy test at screening/pre-first dose. Males planning to father children or unwilling to abstain from sperm donation within 90 days of the last dose of study product.
4. History or presence of clinically relevant (as assessed by the Investigator) cardiovascular, broncho-pulmonary, gastrointestinal, hepatic/ gallbladder*/ bile duct, renal, metabolic, hematological, neurological, musculoskeletal/rheumatological, systemic, ocular, gynaecological, or infectious disease or signs of acute illness. *including medical history of asymptomatic gallbladder stones.
5. Any gastrointestinal surgery or condition or disease that could affect drug absorption, distribution, metabolism or excretion (e.g., gastrectomy, cholecystectomy, diarrhea, recurrent nausea/vomiting).
6. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer considered treated and cured), treated or untreated, within 5 years before screening, regardless of if there is no evidence of local recurrence or metastases.
7. History of schizophrenia, bipolar disorder psychoses, disorders requiring lithium, attempted or planned suicide, or any other severe (disabling) chronic psychiatric diagnosis including depression, generalised anxiety and obsessive-compulsive disorders. Hospitalization within 5 years before screening due to psychiatric illness or due to danger to self or others.
8. Severe recurring headache (cluster or migrainous headaches) requiring prescription medication.
9. Donation of >450 mL blood or blood products within 8 weeks before first dose.
10. Documented evidence of current or past cardiovascular disease including cardiac arrhythmias, clinical significant abnormal cardiac automaticity, or family history of congenital long QT syndrome, Brugada syndrome, or unexplained sudden cardiac death.
11. History or presence of diagnosed (by an allergist/immunologist) or treated (by a physician) food or known drug allergy, or any history of anaphylaxis or other severe allergic reactions including face, mouth, or throat swelling or any difficulty breathing. Allergy, hypersensitivity or intolerance to KS101, including excipients, or to medicinal products with similar chemical structures. Note: Seasonal allergies ('hay fever') or allergy to animal or house dust mite that are untreated and asymptomatic at time of dosing are not exclusionary.
12. Positive serology test at Screening for hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibody, or human immune deficiency virus (HIV) antibody.
13. History of convulsion (including drug or vaccine-induced episodes). Note: Medical history of a single febrile convulsion during childhood is not exclusionary.
14. History of alcohol or illicit drug misuse within 2 years before Screening, as determined by the Investigator and/or positive urine drug test at Screening or pre-first dose (unless there is an explanation deemed acceptable by the Investigator [e.g., false positive] and/or the participant tests negative upon re-test [one re-test permitted per scheduled timepoint]) and/or positive alcohol breath test at Screening or pre-first dose (no re-test permitted).
15. Current tobacco smoker or other nicotine use >5 cigarettes or nicotine equivalent per month within 32 months of Screening, or at Screening or upon admission to the clinical unit had urine cotinine of ≥500 ng/mL or CO breath test >10 ppm.
16. Use of prescription medicines, over-the-counter (OTC) medications (including vitamins), or herbal remedies within 14 days and/or vaccination within 28 days before Day -1. Contraceptives and occasional/non-chronic use (as judged by the Investigator) of non-prescription analgesia (e.g., ibuprofen, paracetamol) are permitted.
17. In the judgement of the Investigator, individual is likely to be noncompliant or unable to comply with study requirements during the study for any reason (e.g., inability to return for follow-up visits, uncooperative attitude), and/or has a medical condition jeopardizing involvement in the study. For Part 2 FE, this includes individuals unwilling or unable to consume a high-fat meal within 30 minutes.
18. Administered an investigational drug within 90 days before first dose, or within 5 times the half-life of the other investigational product (if known), whichever is longer, or previously received study treatment in this study
19. Is vegan.
20. Not willing or able to avoid consumption of grapefruit or Seville oranges or their juices and/or coffee/caffeine-containing beverages within 48 hours before admission to the clinical unit and until discharge from the unit.
21. Identified as a site employee of the Investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that Investigator or study centre, as well as family members (i.e., immediate, husband, wife or de facto and their children, adopted or natural) of the site employees or the Investigator.
22. Considered vulnerable, defined as individuals whose willingness to participate in a clinical study may have been unduly influenced by expectation of benefits associated with participation (justified or not), or of a retaliatory response from senior hierarchy members in case of refusal to participate (e.g., persons in detention, minors, and those incapable of giving informed consent).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of single and multiple ascending oral doses of KS101 in healthy adult volunteers. | Through to end of study, up to 63 days.
  Number of participants reporting treatment emergent adverse events (TEAEs) including treatment-related TEAEs, serious adverse events (SAEs) and TEAEs of severity grade 3 or above.
Evaluation of the safety and tolerability of a single oral dose of KS101 taken after a high-fat meal, assessed by changes observed during the physical examination. | Through to end of study, up to 63 days.
  Presence of clinically significant changes in participants physical examinations post-first dose.
Evaluation of the safety and tolerability of a single oral dose of KS101 taken after a high-fat meal, assessed by changes in haematology parameters. | Through to end of study, up to 63 days.
  Presence of clinically significant changes in participants haematology parameters post-first dose.
Evaluation of the safety and tolerability of a single oral dose of KS101 taken after a high-fat meal, assessed by changes in serum biochemistry. | Through to end of study, up to 63 days.
  Presence of clinically significant changes in participants serum biochemistry parameters post-first dose.
Evaluation of the safety and tolerability of a single oral dose of KS101 taken after a high-fat meal, assessed by changes in coagulation parameters. | Through to end of study, up to 63 days.
  Presence of clinically significant changes in participants coagulation parameters post-first dose.
Evaluation of the safety and tolerability of a single oral dose of KS101 taken after a high-fat meal, assessed by changes in urinalysis parameters. | Through to end of study, up to 63 days.
  Presence of clinically significant changes in participants urinalysis parameters post-first dose.
Evaluation of the safety and tolerability of a single oral dose of KS101 taken after a high-fat meal, assessed by changes in vital signs. | Through to end of study, up to 63 days.
  Presence of clinically significant changes in participants vital signs post-first dose.
Evaluation of the safety and tolerability of a single oral dose of KS101 taken after a high-fat meal, assessed by changes in ECG parameters. | Through to end of study, up to 63 days.
  Presence of clinically significant changes in participants ECG parameters post-first dose.

SECONDARY OUTCOMES:
Pharmacokinetics parameter - High-fat, high-calorie meal effects maximum observed concentration (Cmax). | Through to 7 days post last dose.
  The effect of a standardised high-fat, high-calorie meal on the maximum observed concentration of the study drug in serum will be analyzed for all participants.
Pharmacokinetics parameter - High-fat, high-calorie meal effects on Area under the curve (AUC). | Through to 7 days post last dose.
  The effect of a standardised high-fat, high-calorie meal on the area under the curve of the study drug in serum will be analyzed for all participants.
Pharmacokinetics parameter - High-fat, high-calorie meal effects on time for maximum observed Concentration (Tmax). | Through to 7 days post last dose.
  The effect of a standardised high-fat, high-calorie meal on the Serum PK Tmax will be analyzed for all participants.
Pharmacokinetics parameter - single dose of KS101 effects maximum observed concentration (Cmax). | Through to 7 days post last dose.
  The effect of a single dose of KS101 on the maximum observed concentration of the study drug in serum will be analyzed for all participants.
Pharmacokinetics parameter - multiple doses of KS101 effects maximum observed concentration (Cmax). | Through to 7 days post last dose.
  The effect of multiple doses of KS101 on the maximum observed concentration of the study drug in serum will be analyzed for all participants.
Pharmacokinetics parameter - single dose of KS101 effects on Area under the curve (AUC). | Through to 7 days post last dose.
  The effect of a single dose of KS101 on the area under the curve of the study drug in serum will be analyzed for all participants.
Pharmacokinetics parameter - multiple doses of KS101 effects on Area under the curve (AUC). | Through to 7 days post last dose.
  The effect of multiple doses of KS101 on the area under the curve of the study drug in serum will be analyzed for all participants.
Pharmacokinetics parameter - single dose of KS101 effects on time for maximum observed Concentration (Tmax). | Through to 7 days post last dose.
  The effect of a single dose of KS101 on the Serum PK Tmax will be analyzed for all participants.
Pharmacokinetics parameter - multiple doses of KS101 effects on time for maximum observed Concentration (Tmax). | Through to 7 days post last dose.
  The effect of multiple doses of KS101 on the Serum PK Tmax will be analyzed for all participants.
Pharmacokinetics parameter - single dose of KS101 effects on KS101 half-life (t1/2). | Through to 7 days post last dose.
  The effect of a single dose of KS101 on the KS101 half-life (t1/2) will be analyzed for all participants.
Pharmacokinetics parameter - multiple doses of KS101 effects on KS101 half-life (t1/2) | Through to 7 days post last dose.
  The effect of multiple doses of KS101 on KS101 half-life (t1/2) will be analyzed for all participants.
Pharmacokinetics parameter - multiple doses of KS101 effects on its bioavailability (CL/F). | Through to 7 days post last dose.
  The effect of multiple doses of KS101 on its bioavailability (CL/F) will be analyzed for all participants.
Pharmacokinetics parameter - single dose of KS101 effects on its bioavailability (CL/F). | Through to 7 days post last dose.
  The effect of a single dose of KS101 on its bioavailability (CL/F) will be analyzed for all participants.
Pharmacokinetics parameter - multiple doses of KS101 effects on the apparent volume of distribution (Vz/F). | Through to 7 days post last dose.
  The effect of multiple doses of KS101 on the apparent volume of distribution (Vz/F) will be analyzed for all participants.
Pharmacokinetics parameter - single dose of KS101 effects on the apparent volume of distribution (Vz/F). | Through to 7 days post last dose.
  The effect of a single dose of KS101 on the apparent volume of distribution (Vz/F) will be analyzed for all participants.
Pharmacokinetics parameter - multiple doses of KS101 effects on the apparent elimination rate constant (KEL). | Through to 7 days post last dose.
  The effect of multiple doses of KS101 on the elimination rate constant (KEL) will be analyzed for all participants.
Pharmacokinetics parameter - single dose of KS101 effects on the elimination rate constant (KEL). | Through to 7 days post last dose.
  The effect of a single dose of KS101 on the elimination rate constant (KEL) will be analyzed for all participants.
Pharmacokinetics parameter - multiple doses of KS101 effects on the accumulation index (RAC). | Through to 7 days post last dose.
  The effect of multiple doses of KS101 on the accumulation index (RAC) will be analyzed for all participants.
Investigate the dose proportionality of multiple doses of KS101 on untransformed Cmax. | Through to Day 5.
  For each Part 3 dose: untransformed Cmax will be analysed for all participants.
Investigate the dose proportionality of multiple doses of KS101 on area under the curve (AUC). | Through to Day 5.
  For each Part 3 dose: area under the curve (AUC) will be analysed for all participants.
investigate the dose proportionality of single doses of KS101 on untransformed CMAX. | Through to end of study, up to 63 days.
  For each Part 1 dose: untransformed Cmax will be analysed for all participants.
investigate the dose proportionality of single doses of KS101 on the area under the curve (AUC). | Through to end of study, up to 63 days.
  For each Part 1 dose: the area under the curve (AUC) will be analysed for all participants.

OTHER OUTCOMES:
Characterize the PK profile of KS101 in the urine of healthy adult participants after single ascending oral doses of KS101. | Through to 24 hours post KS101 dose.
  Estimation of KS101 PK parameters after single dose including, but not limited to, Ae0-24, Fe0-24, CLr.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No